CLINICAL TRIAL: NCT05460949
Title: Effects of William Training Versus Hold Relax Stretching of Iliopsoas Muscle in Females With Hyperlordosis
Brief Title: William Training Versus Hold Relax Stretching of Iliopsoas Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0520
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Hyperlordosis
MeSH Terms: conditions — Swayback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOLD RELAX STRETCHING OF ILIOPSOAS (Experimental): 10-second isometric contraction of iliopsoas muscle (HR), 10-second rest, 20-second static stretch, 5 repetitions.
  The stretching exercise was performed 2 times a week for 8 weeks.
  Interventions: Other: HOLD RELAX STRETCHING OF ILIOPSOAS
- • WILLIAM'S PROTOCOL (Experimental): * Pelvic tilt
  * Single Knee to chest
  * Double knee to chest
  * Partial sit-up
  * Hamstring stretch
  * Hip Flexor stretch
  * Squat
  * Each group performed special trainings for 8 weeks, 2 sessions per week; each session took about 1 hour. Duration of each exercise was 8 to 10 seconds in each set. Protocols were started with 1 set of 10 repetitions at starting baseline and by improving performance and patients' compatibility with trainings, all eventually finished with 3 sets of 20 repetitions at the end of protocols.
  Interventions: Other: WILLIAM'S PROTOCOL

INTERVENTIONS:
Other: HOLD RELAX STRETCHING OF ILIOPSOAS — 10 second isometric contraction of iliopsoas muscle (HR), 10-second rest, 20 second static stretch, 5 repetitions.
  • The stretching exercise was performed 2 times a week for 8 weeks. 10 second isometric contraction of iliopsoas muscle (HR), 10-second rest, 20 second static stretch, 5 repetitions.
  The stretching exercise was performed 2 times a week for 8 weeks.
  Arms: HOLD RELAX STRETCHING OF ILIOPSOAS
Other: WILLIAM'S PROTOCOL — Pelvic tilt Single Knee to chest Double knee to chest Partial sit-up Hamstring stretch Hip Flexor stretch Squat Each group performed special trainings for 8 weeks, 2 sessions per week; each session took about 1 hour. Duration of each exercise was 8 to 10 seconds in each set. Protocols were started with 1 set of 10 repetitions at starting baseline and by improving performance and patients' compatibility with trainings, all eventually finished with 3 sets of 20 repetitions at the end of protocols.
  Arms: • WILLIAM'S PROTOCOL

SUMMARY:
Hyper lordosis is a condition in which there is an excessive spine curvature in the lower back. Hyper lordosis is a very common symptom. It occurs in high-income, middle-income, and low-income countries and all age groups from children to the elderly population Only a small proportion of people have a well understood pathological cause-eg, a vertebral fracture, malignancy, or infection. People with physically demanding jobs, physical and mental comorbidities, smokers, and obese individuals are at greatest risk of reporting low back pain.Hyper lordosis creates a characteristic C-shaped curve in the lower back, or lumbar region, where the spine curves inward just above the buttocks. It often occurs as a result of poor posture or a lack of exercise. Hyperlordosis can cause muscle tightening and stiffness in the lower back. It can also damage the spine and soft tissues in the lumbar region. Hyperlordosis leads to excessive curvature of the spine in the lower back, causing the abdomen and buttocks to appear more prominent in profile view. People with hyperlordosis may experience mild to severe lower back pain, which may worsen with movement.

Various conservative treatments are used to treat hyperlordosis and low back pain due to hyperlordosis. Most commonly used are the manual therapy techniques that employ William's protocol and hold relax stretching of iliopsoas muscle at lumbar spine. This study will be randomized control trial used to compare the effects of William protocol and hold relax stretching of iliopsoas muscle in subjects with hyperlordosis and low back pain. Subjects meeting the predetermined inclusion and exclusion criteria will be divided into two groups using lottery method. Pre assessment will be done using LUMBAR SPINE QUESTIONNAIRE as subjective measurements and NPRS as objective measurements. Subjects in one group will be treated using William's protocol and the other one will be treated with hold relax stretching of iliopsoas muscle. Each subject will receive 08 treatment sessions with 02 treatment sessions per week. Post treatment reading for NPRS and lumbar spine questionnaire will be recorded after every week.

DETAILED DESCRIPTION:
Hyper lordosis is a condition in which there is an excessive spine curvature in the lower back. Hyper lordosis is a very common symptom. It occurs in high-income, middle-income, and low-income countries and all age groups from children to the elderly population Only a small proportion of people have a well understood pathological cause-eg, a vertebral fracture, malignancy, or infection. People with physically demanding jobs, physical and mental comorbidities, smokers, and obese individuals are at greatest risk of reporting low back pain.Hyper lordosis creates a characteristic C-shaped curve in the lower back, or lumbar region, where the spine curves inward just above the buttocks. It often occurs as a result of poor posture or a lack of exercise. Hyperlordosis can cause muscle tightening and stiffness in the lower back. It can also damage the spine and soft tissues in the lumbar region. Hyperlordosis leads to excessive curvature of the spine in the lower back, causing the abdomen and buttocks to appear more prominent in profile view. People with hyperlordosis may experience mild to severe lower back pain, which may worsen with movement.

Various conservative treatments are used to treat hyperlordosis and low back pain due to hyperlordosis. Most commonly used are the manual therapy techniques that employ William's protocol and hold relax stretching of iliopsoas muscle at lumbar spine. This study will be randomized control trial used to compare the effects of William protocol and hold relax stretching of iliopsoas muscle in subjects with hyperlordosis and low back pain. Subjects meeting the predetermined inclusion and exclusion criteria will be divided into two groups using lottery method. Pre assessment will be done using LUMBAR SPINE QUESTIONNAIRE as subjective measurements and NPRS as objective measurements. Subjects in one group will be treated using William's protocol and the other one will be treated with hold relax stretching of iliopsoas muscle. Each subject will receive 08 treatment sessions with 02 treatment sessions per week. Post treatment reading for NPRS and lumbar spine questionnaire will be recorded after every week.Various conservative treatments are used to treat hyperlordosis and low back pain due to hyperlordosis. Most commonly used are the manual therapy techniques that employ William's protocol and hold relax stretching of iliopsoas muscle at lumbar spine. This study will be randomized control trial used to compare the effects of William protocol and hold relax stretching of iliopsoas muscle in subjects with hyperlordosis and low back pain. Subjects meeting the predetermined inclusion and exclusion criteria will be divided into two groups using lottery method. Pre assessment will be done using LUMBAR SPINE QUESTIONNAIRE as subjective measurements and NPRS as objective measurements. Subjects in one group will be treated using William's protocol and the other one will be treated with hold relax stretching of iliopsoas muscle. Each subject will receive 08 treatment sessions with 02 treatment sessions per week. Post treatment reading for NPRS and lumbar spine questionnaire will be recorded after every week.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-40 years
* Hyperlordosis Angle
* Females having increased lordotic curve
* Pain perceived anywhere in the region of lumbar spine from L1 to l5.
* Limitation of lumbar spine range of motion.

Exclusion Criteria:

* Any red flags including tumors, fractures.
* Spinal canal stenosis
* Rheumatoid arthritis
* Osteoporosis

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
pain assessment | 8 weeks
  The NRS for pain is a unidimensional measure of pain intensity in adults including those with chronic pain due to rheumatic diseases. Although various iterations exist, the most commonly used is the 11-item NRS
lordatic angle | 8 weeks
  2- Flexicurve ruler: The angle of lumbar lordosis will be measured with a flexible ruler. The subject remained in the normal standing posture while lordatic angle was measured
low back pain | 8 weeks
  3- Lumbar spine questionnaire (LSQ): It is used for the assessment of low back pain. It contains various items and patients will be asked relevant questions and answers will be noted and written

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, MSWHPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No